CLINICAL TRIAL: NCT07344116
Title: Establishment of a Hepatobiliary and Pancreatic Tumor Biobank at a Single Academic Medical Center
Brief Title: Hepatobiliary and Pancreatic Tumor Biobank
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, jinyun, PhD, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: ZJU2-HBP-BIOBANK-LJT
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hepotacellular Carcinoma; Cholangiocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatobiliary and Pancreatic Biobank Participants: Participants enrolled in this observational biobank study, including patients with hepatobiliary and pancreatic malignant tumors, patients with benign hepatobiliary and pancreatic diseases, and selected healthy volunteers. Biological specimens and related clinical data are collected during routine clinical care without experimental interventions.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — This is an observational biobank study. No experimental intervention, treatment, or procedure is assigned as part of the study. Biological specimens are collected only during routine clinical care or from remaining clinical specimens.

SUMMARY:
This study aims to establish a hepatobiliary and pancreatic tumor biobank at the Second Affiliated Hospital of Zhejiang University School of Medicine. The biobank will systematically collect and store human biological samples, such as blood, tissue, bile, and other body fluids, together with relevant clinical and follow-up information from patients with hepatobiliary and pancreatic tumors, benign hepatobiliary and pancreatic diseases, and selected healthy volunteers.

The collection of samples will be performed without changing routine medical care and will not involve any experimental treatment or additional invasive procedures for research purposes. Biological samples will be obtained during standard clinical diagnosis and treatment, or from remaining specimens after routine clinical use.

All samples and data will be coded and stored according to ethical and legal requirements to protect participants' privacy. The biobank is intended to serve as a long-term research resource to support future basic, translational, and clinical research on hepatobiliary and pancreatic diseases, with the goal of improving understanding of disease mechanisms and advancing medical research in this field.

DETAILED DESCRIPTION:
This study is designed as a single-center, observational biobank project conducted at the Second Affiliated Hospital of Zhejiang University School of Medicine. The primary purpose of this study is to establish and maintain a structured hepatobiliary and pancreatic tumor biobank that integrates biological specimens with corresponding clinical and follow-up data for long-term research use.

Eligible participants include adult patients diagnosed with hepatobiliary and pancreatic malignant tumors, patients with benign hepatobiliary and pancreatic diseases, and selected healthy volunteers. Enrollment is based on predefined inclusion and exclusion criteria, and participation requires written informed consent unless otherwise approved by the institutional ethics committee for retrospective samples.

Biological specimens collected in this biobank may include peripheral blood, tumor and adjacent non-tumor tissue, bile, and other body fluids. Sample collection is performed without altering routine medical care and does not involve experimental treatments or additional invasive procedures for research purposes. Specimens are obtained during standard diagnostic or therapeutic procedures or from remaining clinical specimens after routine use.

Clinical information associated with each participant, such as demographic characteristics, diagnosis, pathology findings, treatment details, and follow-up outcomes, is systematically collected from existing medical records and follow-up systems. All data and specimens are coded and de-identified prior to storage to ensure participant confidentiality.

The biobank is intended to function as a long-term research infrastructure. Biological samples and data may be used in future ethically approved basic, translational, or clinical studies related to hepatobiliary and pancreatic diseases. Each secondary use of samples or data will require appropriate ethical review and approval in accordance with institutional and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients diagnosed with hepatobiliary or pancreatic malignant tumors, including but not limited to hepatocellular carcinoma, cholangiocarcinoma, gallbladder cancer, and pancreatic cancer; or patients with benign hepatobiliary or pancreatic diseases; or selected healthy volunteers.
* Receiving medical care or health evaluation at the Second Affiliated Hospital of Zhejiang University School of Medicine.
* Able and willing to provide written informed consent, unless waived or exempted by the institutional ethics committee for retrospective samples.
* Willing to allow collection and storage of biological specimens and related clinical data for research purposes.

Exclusion Criteria:

* Age younger than 18 years.
* Unable to provide informed consent and without a legally authorized representative.
* Presence of conditions that, in the opinion of the investigators, make participation inappropriate or infeasible.
* Refusal to allow the collection or use of biological specimens or clinical data for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients receiving care at the Second Affiliated Hospital of Zhejiang University School of Medicine who are diagnosed with hepatobiliary or pancreatic malignant tumors, as well as patients with benign hepatobiliary or pancreatic diseases. Selected healthy adult volunteers may also be included as controls. Participants are enrolled without altering routine medical care, and biological specimens and related clinical data are collected for biobanking and future research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2036-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful Establishment of a Hepatobiliary and Pancreatic Tumor Biobank | up to 5 years

IPD SHARING:
Plan to Share IPD: No